CLINICAL TRIAL: NCT03757364
Title: Effect of Methotrexate in the Treatment of Distal Interphalangeal Joint Extensor Tendon Enthesopathy in Patients With Nail Psoriasis
Brief Title: Methotrexate in the Treatment of Distal Interphalangeal Joint Extensor Tendon Enthesopathy in Nail Psoriasis
Status: Completed | Type: Observational
Sponsor: Ryszard Górecki (Other)
Responsible Party: Sponsor-Investigator, Ryszard Górecki, Head of Collegium Medicum, Clinical Professor, University of Warmia and Mazury
Organization: University of Warmia and Mazury (Other)
Other Study IDs: UWM/Ps-ENTH.2018/001
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Nail Psoriasis
Keywords: Distal Interphalangeal Joint Extensor Tendon Enthesopathy; Nail Psoriasis
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood probes for laboratory test
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 19 patients with Ps: 19 patients with Ps with psoriatic changes in nails treated at the Dermatological Clinic in Olsztyn and the Clinic of Dermatology, Sexually Transmitted Diseases and Clinical Immunology of the University of Warmia and Mazury in Olsztyn, in whom a US examination revealed DIP joint extensor tendon enthesopathy who were started on methotrexate during the study and the treatment continued for 6 months
  Interventions: Drug: Methotrexate
- 13 patients with PsA: 13 patients with PsA with psoriatic changes in nails treated at the Dermatological Clinic in Olsztyn and the Clinic of Dermatology, Sexually Transmitted Diseases and Clinical Immunology of the University of Warmia and Mazury in Olsztyn, in whom a US examination revealed DIP joint extensor tendon enthesopathy who were started on methotrexate during the study and the treatment continued for 6 months
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Methotrexate in the treatment of distal interphalangeal joint extensor tendon enthesopathy in patients with nail psoriasis
  Other Names: Methotrexate Ebeve, Metex,

SUMMARY:
The primary aim of the study is to assess the effect of methotrexate on the development of distal interphalangeal joint extensor tendon enthesopathy.

DETAILED DESCRIPTION:
Nail psoriasis is one of the risk factors for psoriatic arthritis (PsA), especially with distal interphalangeal joints affected. Nail changes in psoriasis have been observed in 10-55% of patients, and the nail psoriasis-related inflammation can spread to adjacent structures, including DIP joints and digital extensor tendons. Enthesopathies are among the characteristic features of psoriatic arthritis. In everyday practice, assessment of psoriatic changes in nails is based mainly on clinical indices, such as nail psoriasis severity index (NAPSI) and modified NAPSI (mNAPSI), while imaging examinations, such as ultrasonography are performed much less frequently.

The findings of this study may assess the reasonableness of systemic treatment of nail psoriasis in patients without arthritis as enthesopathy prevention as well as the usability of US nail examinations in Ps and PsA patients in assessment of morphological changes and a response to treatment.

A US examination of nails and distal interphalangeal joint extensor tendons are conducted in all of the patients twice at an interval of six months. The examination is conducted by a rheumatologist experienced in ultrasound examinations of the skeletal and muscular system. An assessment of the nails, extensor tendons and DIP joints is made by placing the head on the dorsal side. In order to avoid pressure on surface tissues, an appropriate amount of gel without gel pads was used. The intensified blood flow, made visible by the PD technique, is confirmed by pulsed wave Doppler spectrum. The nail thickness is measured as the maximum distance between the dorsal and ventral nail plates. The nail bed thickness is measured as the distance between the ventral plate and the bone margin of the distal phalanx. The nail matrix thickness is measured at the proximal end of the nail bed.

The study was approved by the Bioethics Committee of the Warmia and Mazury Chamber of Physicians The study are conducted according to the Good Clinical Practice guidelines. Each participant signs an informed consent and be coded with unique ID.

Results of analyses will be saved by indexing with ID code only, personal data with individual IDs will be saved in additional file. All hard copy will be archived in secure room with coded electronic key.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriatic changes in nails treated at the Rheumatological Clinic in Olsztyn and the Clinic of Dermatology, Sexually Transmitted Diseases and Clinical Immunology of the University of Warmia and Mazury in Olsztyn, in whom a US examination revealed DIP joint extensor tendon enthesopathy

Exclusion Criteria:

* Patients diagnosed with osteoarthritis of hands, those who work hard physically and those with changes in nails other than caused by psoriasis

Ages: 34 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with psoriatic changes in nails with distal interphalangeal extensor tendon enthesopathy in ultrasound examination
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Effect of Methotrexate on Distal Interphalangeal Joint Extensor Tendon Enthesopathy | 6 months
  Ultrasonographic assessment of the effect of methotrexate on the development of distal interphalangeal joint extensor tendon enthesopathy in patients with nail psoriasis.

SECONDARY OUTCOMES:
Effect of Methotrexate on Morphological Changes in Psoriatic Nails | 6 months
  Ultrasonographic assessment of the effect of methotrexate on morphological changes in psoriatic nails

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Krajewska-Włodarczyk, PhD, Principal Investigator — University of Warmia and Mazury
Locations (1):
- University of Warmia and Mazury, Olsztyn, Warmian-Masurian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krajewska-Wlodarczyk M, Owczarczyk-Saczonek A, Placek W, Wojtkiewicz M, Wiktorowicz A, Wojtkiewicz J. Ultrasound Assessment of Changes in Nails in Psoriasis and Psoriatic Arthritis. Biomed Res Int. 2018 Sep 9;2018:8251097. doi: 10.1155/2018/8251097. eCollection 2018. PMID 30271786
- [Background] McGonagle D, Tan AL, Benjamin M. The nail as a musculoskeletal appendage--implications for an improved understanding of the link between psoriasis and arthritis. Dermatology. 2009;218(2):97-102. doi: 10.1159/000182250. Epub 2008 Dec 6. PMID 19060455
- See also: Ultrasound Assessment of Changes in Nails in Psoriasis and Psoriatic Arthritis — https://www.ncbi.nlm.nih.gov/pubmed/30271786
- See also: The link between psoriasis and arthritis — https://www.ncbi.nlm.nih.gov/pubmed/19060455